CLINICAL TRIAL: NCT07330063
Title: Efficacy and Safety of Anrikefon Injection for the Treatment of Postoperative Pain in Patients Undergoing Totally Laparoscopic Radical Distal Gastrectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E20251321
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Gastrectomy
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Normal Saline via intravenous bolus injection, once every 8 hours (q8h), for a total of 6 doses.
  Interventions: Drug: Placebo Group
- Anruikfen Intravenous Bolus Injection Group (Experimental): Anruikefen 1 μg/kg via intravenous bolus injection, once every 8 hours (q8h), for a total of 6 doses.
  Interventions: Drug: Anruikefen (Intravenous Bolus)
- Anruikefen Intravenous Infusion Group (Experimental): Anruikefen 1.5 μg/kg via intravenous infusion, once every 8 hours (q8h), for a total of 6 doses.
  Interventions: Drug: Anruikefen (Intravenous Infusion)

INTERVENTIONS:
Drug: Anruikefen (Intravenous Bolus) — Anruikefen 1 μg/kg via intravenous bolus injection, once every 8 hours (q8h), for a total of 6 doses.
  Arms: Anruikfen Intravenous Bolus Injection Group
Drug: Anruikefen (Intravenous Infusion) — Anruikefen 1.5 μg/kg via intravenous infusion, once every 8 hours (q8h), for a total of 6 doses.
  Arms: Anruikefen Intravenous Infusion Group
Drug: Placebo Group — Normal Saline administered via intravenous bolus injection, once every 8 hours (q8h), for a total of 6 doses.
  Arms: Placebo Group

SUMMARY:
Anruikefen is a peripherally highly selective kappa receptor agonist that does not easily cross the blood-brain barrier, resulting in a low incidence of central adverse reactions such as respiratory depression, sedation, and addiction. As a Class 1 new drug, it was approved for marketing in China on May 13, 2025, and is indicated for the treatment of postoperative pain following abdominal surgery. Results from two Phase Ⅲ randomized controlled trials (RCTs) of Anruikefen have demonstrated its significant analgesic efficacy, with the incidence of postoperative nausea and vomiting (PONV) being 50% significantly lower than that in the placebo group, which confirms the favorable safety profile of Anruikefen Injection.

Therefore, this investigator-initiated trial (IIT) is designed to further verify the efficacy and safety of Anruikefen in patients undergoing total laparoscopic distal gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old (inclusive).
* American Society of Anesthesiologists (ASA) physical status classification Class I-III.
* Body Mass Index (BMI) ranging from 18 kg/m² to 30 kg/m² (inclusive).
* Patients scheduled for elective total laparoscopic distal gastrectomy for gastric cancer under general anesthesia, with surgical duration < 5 hours.
* Surgical incision length < 8 cm.
* Voluntarily agree to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Patients undergoing emergency surgery or suffering from trauma.
* Patients who undergo conversion to open surgery or laparoscopically assisted distal gastrectomy for gastric cancer during the operation.
* Patients who refuse to receive Patient-Controlled Intravenous Analgesia (PCIA).
* Patients with a history of prior abdominal surgery.
* Patients expected to require prolonged endotracheal intubation after surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Consumption of Sufentanil via PCIA | within 48 Hours after the First Administration Postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, 不限, China

IPD SHARING:
Plan to Share IPD: Undecided